CLINICAL TRIAL: NCT00294879
Title: Effects of Inspiration Rise Time on Work of Breathing and Comfort of Conscious Patients on Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Radboud University Nijmegen Medical Centre, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: LBCH 0601
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Mechanical Ventilation

INTERVENTIONS:
Procedure: pressure support ventilation at 0, 5, and 10% IRT

SUMMARY:
Introduction Pressure Support Ventilation is widely used in patients in the ICU. Matching the patient's respiratory needs with adequate ventilator settings is necessary to ensure a low work of breathing (WOB) and maximal patient comfort. The inspiratory rise time (IRT) determines the time to reach the selected airway pressure. A short IRT results in a high peak inspiratory flow and a short time to reach that peak, but is also associated with the development of turbulent flow, resulting in increased WOB. Aim of this study is to investigate the effects of different IRT settings on WOB and patient comfort during pressure support ventilation.

Methods We will performed a prospective, single blind cohort study in patients on Pressure Support Ventilation. 10 healthy adult patients admitted to the ICU after elective facial or neck surgery will be included. All patients will be ventilated in pressure support mode using a Servo 300 ventilator (Siemens. Elema, Solna, Sweden), with a positive end expiratory pressure of 5 cm H2O, pressure support level of 12 cm H2O above PEEP and an inspiratory oxygen fraction of 0.40. Patients have to be awake and cooperative (Ramsay 2). WOB will be measured with an esophageal balloon, and miniature flowmeter (Bicore system). Breathing comfort will be evaluated using a visual analogue scale (VAS) ranging from 1 to 10. WOB and patient comfort will be measured (in random order) at 0, 5, and 10% IRT. For statistical analysis the two-way analysis of variance will used. A p value of < 0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
Introduction Pressure Support Ventilation is widely used in patients in the ICU. Matching the patient's respiratory needs with adequate ventilator settings is necessary to ensure a low work of breathing (WOB) and maximal patient comfort. The inspiratory rise time (IRT) determines the time to reach the selected airway pressure. A short IRT results in a high peak inspiratory flow and a short time to reach that peak, but is also associated with the development of turbulent flow, resulting in increased WOB. Aim of this study is to investigate the effects of different IRT settings on WOB and patient comfort during pressure support ventilation.

Methods We will performed a prospective, single blind cohort study in patients on Pressure Support Ventilation. 10 healthy adult patients admitted to the ICU after elective facial or neck surgery will be included. All patients will be ventilated in pressure support mode using a Servo 300 ventilator (Siemens. Elema, Solna, Sweden), with a positive end expiratory pressure of 5 cm H2O, pressure support level of 12 cm H2O above PEEP and an inspiratory oxygen fraction of 0.40. Patients have to be awake and cooperative (Ramsay 2). WOB will be measured with an esophageal balloon, and miniature flowmeter (Bicore system). Breathing comfort will be evaluated using a visual analogue scale (VAS) ranging from 1 to 10. WOB and patient comfort will be measured (in random order) at 0, 5, and 10% IRT. For statistical analysis the two-way analysis of variance will used. A p value of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* awake and cooperative patient
* ICU admission following surgery of head or neck

Exclusion Criteria:

* coagulopathy
* inability to sit
* hypoxemia and/or hypercapnia and /or hypocapnia
* Pain score > 5 (on scale 1-10)
* esophageal abnormalities
* Pregnancy
* COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-02; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Work of breathing

SECONDARY OUTCOMES:
patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia WE Hoedemaekers, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands